CLINICAL TRIAL: NCT00805350
Title: Efficacy and Safety of Eplivanserin 5mg/Day in Insomnia Characterized by Sleep Maintenance Difficulties: a 6-week, Randomized, Double-blind, Placebo-controlled, Polysomnography Study.
Brief Title: Efficacy and Safety of Eplivanserin 5mg/Day in Insomnia Characterized by Sleep Maintenance Difficulties
Acronym: ECLIPSE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EFC10844; 2008-003791-22 (EudraCT Number)
Record Dates: First submitted 2008-12-04; First posted 2008-12-09 (Estimated); Last update posted 2016-03-07 (Estimated); Status verified 2016-02

CONDITIONS: Primary Insomnia
Keywords: Insomnia; Sleep Maintenance; Polysomnography
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — SR 46349B

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Eplivanserin (Experimental): Eplivanserin 5 mg/day
  Interventions: Drug: Eplivanserin
- Placebo (Placebo Comparator): Placebo of Eplivanserin 5 mg/day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Eplivanserin — one 5 mg tablet once a day
  Other Names: SR46349
  Arms: Eplivanserin
Drug: Placebo — Placebo of Eplivanserin one tablet once a day
  Arms: Placebo

SUMMARY:
Primary objective:

- To assess the efficacy of eplivanserin 5mg/day in comparison to placebo after 6 weeks of treatment on sleep maintenance of insomniac patients, as measured by Polysomnography Wake Time After Sleep Onset (PSG-WASO) and Polysomnography Number of Awakenings (PSG-NAW).

Secondary objectives:

* To evaluate the effects of eplivanserin 5mg/day as compared to placebo after 6 weeks of treatment on other sleep parameters measured by PSG recordings (Total Sleep Time - PSG-TST, Sleep Efficiency - PSG-SE, Latency to Persistent Sleep - PSG-LPS) and reported by patients (Wake Time After Sleep Onset - pr-WASO, Number of Awakenings - pr-NAW, Total Sleep Time - pr-TST, Quality of Sleep - QoS and Refreshing Quality of Sleep - RqoS).
* To evaluate the effects of eplivanserin 5mg/day on sleep architecture compared to placebo.
* To evaluate the effect of eplivanserin 5mg/day on daytime functioning using the Sleep Impact Scale (SIS), as compared with placebo after 6 weeks of treatment.
* To evaluate patient's impression of treatment effects using the Patient's Global Impression questionnaire.
* To evaluate the potential for next-day residual effects (using patient's morning questionnaire and psychometric tests) with eplivanserin 5mg/day as compared to placebo.
* To evaluate the potential for rebound insomnia following abrupt discontinuation of eplivanserin 5mg/day in comparison with placebo.
* To evaluate the effect of eplivanserin, compared to placebo, on the quality of life of patients with primary insomnia using the SF-36 Health Survey.
* To evaluate the clinical safety and tolerability of eplivanserin 5mg/day compared to placebo.

DETAILED DESCRIPTION:
Randomized, double-blind, placebo, controlled study with 2 parallel groups Duration of treatment : 6 weeks

Duration of observation: 9 weeks

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary insomnia based on DSM-IV-TR (Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition - Text Revisions) criteria

Exclusion Criteria:

* Inpatients.
* Mean screening PSG-WASO for screening night 1+ screening night 2 < 45 mn, or screening night with PSG-WASO < 30 mn.
* Mean screening PSG-TST for screening night 1 + screening night 2 ≥7 hours or ≤3hours.
* Mean screening PSG-LPS for screening night 1+ screening night 2 > 30 mn.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 637 (Actual)
Dates: Start 2008-12; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline of mean PSG-WASO on N41/N42 | 6 weeks
Change from baseline of mean PSG-NAW on N41/N42 | 6 weeks

SECONDARY OUTCOMES:
Other PSG sleep parameters: PSG-TST, PSG-SE (TST/Time in Bed), PSG-LPS | 6 weeks
Patient-reported sleep parameters | 6 weeks
Patient Global impression (PGI) | 6 weeks
sleep architecture: percentage of time spent in each sleep stage (1, 2, 3-4/SWS, REM), shift to stage 1, shift to wake, stage 1 + WASO, [stages 3&4]/[stage 1 + WASO]). | 6 weeks
Sleep Impact Scale (SIS) | 6 weeks
SF-36 Health Survey | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (7):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States
- Sanofi-Aventis Administrative Office, Vienna, Austria
- Sanofi-Aventis Administrative Office, Laval, Canada
- Sanofi-Aventis Administrative Office, Paris, France
- Sanofi-Aventis Administrative Office, Berlin, Germany
- Sanofi-Aventis Administrative Office, Budapest, Hungary
- Sanofi-Aventis Administrative Office, Warsaw, Poland